CLINICAL TRIAL: NCT04176367
Title: AN OPEN LABEL, RANDOMIZED, SINGLE DOSE, 2 WAY CROSSOVER BIOEQUIVALENCE STUDY COMPARING NICERGOLINE 10 MG TABLET (MANUFACTURED AT PFIZER DALIAN, CHINA) WITH NICERGOLINE 10 MG TABLET (MANUFACTURED AT PFIZER ITALIA S.R.L., ITALY) UNDER FASTED AND FED CONDITIONS IN HEALTHY CHINESE PARTICIPANTS
Brief Title: An Bioequivalence Study Comparing Nicergoline 10 mg Tablet Manufactured in China With Nicergoline 10 mg Tablet Manufactured in Italy Under Fasted and Fed Conditions in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A7921006
Record Dates: First submitted 2019-11-06; First posted 2019-11-25 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2020-11

CONDITIONS: Pharmacokinetics
Keywords: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test: Nicergoline manufactured in China (Experimental)
  Interventions: Drug: Nicergoline from China
- Reference: Nicergoline manufactured in Italy (Active Comparator)
  Interventions: Drug: Nicergoline from Italy

INTERVENTIONS:
Drug: Nicergoline from China — This is the test arm of China local manufactured Nicergoline
  Arms: Test: Nicergoline manufactured in China
Drug: Nicergoline from Italy — This is the reference arm of Italy originator Nicergoline.
  Arms: Reference: Nicergoline manufactured in Italy

SUMMARY:
This trial is a bioequivalence study to support a generic consistency evaluation program, initiated by the China Food and Drug Administration (CFDA) in 2015, for the evaluation of quality and efficacy of the products manufactured in China. Related guidance was issued by Center for Drug Evaluation (CDE) on 27 Nov 2015 named "Use pharmacokinetic (PK) parameter as endpoint for chemical generics bioequivalence (BE) study".

Nicergoline localized product is manufactured at Pfizer Dalian China, while the reference product is manufactured at Pfizer Italia S.r.l., Italy. The selected strength of 10 mg tablet is the marketed strength in China, and the selected dose of 30 mg (3 x 10 mg tablet) is one of the commonly used clinically approved daily doses with good tolerability profile.

In each group, participants will be randomized to one of the 2 treatment sequences according to a computer generated randomization schedule. Each treatment sequence will consist of 2 periods, separated by a washout period of at least 7 days between the first day of each period.

ELIGIBILITY:
Inclusion Criteria:

Age and Sex:

1. Male and female participants must be 18 to 55 years of age, inclusive, at the time of signing the informed consent document (ICD).

   • Refer to Appendix 4 for reproductive criteria for male (Section 10.4.1) and female (Section 10.4.2) participants.

   Type of Participant and Disease Characteristics:
2. Male and female participants who are overtly healthy as determined by medical evaluation including a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate (PR) measurement, chest radiograph (posteroanterior), 12 lead electrocardiogram (ECG), and clinical laboratory tests.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Participants must be of Chinese ethnicity (individuals currently residing in mainland China who were born in China and have both parents of Chinese descent).

   Weight:
5. Body mass index (BMI) of 18 to 28 kg/m2, inclusive; and a total body weight >50 kg for males and >=45 kg for females.

   Informed Consent:
6. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol.

   Other Inclusions:
7. Participants need to be CYP2D6 non-poor metabolizer (which includes EM, IM and UM) as confirmed by genotype (see Section 8.7.1).

Exclusion Criteria:

Medical Conditions:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy, appendectomy).
3. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B surface antibody (HepBsAb); hepatitis B virus e antigen (HepBeAg); hepatitis B virus e antibody (HepBeAb); hepatitis B core antibody (HepBcAb), hepatitis C antibody (HCVAb) or treponema pallidum antibody (TPPA). Hepatitis B vaccination is allowed.
4. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.

   Prior/Concomitant Therapy:
5. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product. (Refer to Section 6.5 for additional details).
6. Taking any medicinal product that changes the activity of hepatic enzymes within 28 days prior to Screening, such as inducer of CYP2D6.

   Prior/Concurrent Clinical Study Experience:
7. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product used in this study (whichever is longer).

   Diagnostic Assessments:
8. A positive urine drug screen.
9. Screening supine blood pressure (BP) >=140 mm Hg (systolic) or >= 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is >= 140 mm Hg (systolic) or >= 90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
10. Baseline 12 lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline corrected QT (QTc) interval >450 millisecond [msec], complete left bundle branch block [LBBB], signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree atrioventricular [AV] block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate corrected using the Fridericia method and the resulting corrected QT (QTcF) should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.

    Other Exclusions:
11. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
12. Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day within 3 months of Screening; a positive urine nicotine test.
13. Blood donation (excluding plasma donations) of approximately 400 mL or more within 60 days prior to dosing.
14. History of sensitivity to heparin or heparin induced thrombocytopenia.
15. History of hypersensitivity to the active substance or to ergot alkaloids, or to any of the excepients.
16. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
17. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
AUCinf of MDL (area under the plasma concentration-time profile derived from plasma from time 0 extrapolated to infinity) | At the end of Day 11
  MDL is the primary metabolizer of Nicergoline
AUClast of MDL (area under the plasma concentration-time profile derived from plasma from time 0 to the last quantifiable concentration) | At the end of Day 11
  MDL is the primary metabolizer of Nicergoline
Cmax of MDL (maximum observed concentration derived from plasma) | At the end of Day 11
  MDL is the primary metabolizer of Nicergoline

SECONDARY OUTCOMES:
AUCinf of MMDL (area under the plasma concentration-time profile derived from plasma from time 0 extrapolated to infinity) | At the end of Day 11
  MMDL is the secondary metabolizer of Nicergoline
AUClast of MMDL (area under the plasma concentration-time profile derived from plasma from time 0 to the last quantifiable concentration) | At the end of Day 11
  MMDL is the secondary metabolizer of Nicergoline
Cmax of MMDL (maximum observed concentration derived from plasma) | At the end of Day 11
  MMDL is the secondary metabolizer of Nicergoline
Percentage of participants with treatment emergent adverse events | At the end of follow-up phone call that takes place 35-42 days after last study dose (total period of approximately 70 days)
Percentage of participants with clinical laboratory test results above/below certain threshold | At the end of Day 11
Percentage of participants with vital signs above/below certain threshold | At the end of Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Beijing Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A7921006